CLINICAL TRIAL: NCT06913946
Title: Validity of the 'My Nutrition Index' (MNI) and Its Relationship With the Healthy Eating Index-2015 in the Turkish Population
Brief Title: Validity of MNI and Its Relationship With HEI-2015
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Emine Elibol, Assist. Prof., Ankara Yildirim Beyazıt University
Other Study IDs: AYBUELİBOL0010
Record Dates: First submitted 2025-03-31; First posted 2025-04-06 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-03

CONDITIONS: Healthy People
Keywords: My Nutrition Index, Healthy Eating Index, Dietary Assessment

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- adults: The study included 498 individuals aged 19-65. Data were collected using a demographic survey, Three-Day Food Consumption Record Form, and the International Physical Activity Questionnaire. The Three-Day Food Consumption Record Form was used to calculate the MNI and HEI-2015.

SUMMARY:
This study assessed the validity of the "My Nutrition Index" (MNI) and its relationship with the Healthy Eating Index-2015 (HEI-2015) in the Turkish population. A cross-sectional study of 498 participants aged 19-64 years was conducted, collecting demographic, anthropometric, and three-day food consumption data to calculate both indices. Pearson's correlation was used for analysis.

DETAILED DESCRIPTION:
Introduction: Healthy eating is a crucial concept encompassing biochemical, physical, and psychosocial domains, and various nutritional indices and scales have been developed to assess the healthfulness of individuals' diets.

Objective: This study aimed to evaluate the validity of the "My Nutrition Index" (MNI) and examine its relationship with the Healthy Eating Index-2015 (HEI-2015) in the Turkish population.

Methods: This cross-sectional study included 498 participants aged 19-64 years. Demographic and anthropometric data were collected, and three-day food consumption records were obtained to calculate both the My Nutrition Index and the Healthy Eating Index-2015. Participants' nutritional data were analyzed, and the relationship between the two indices was examined using Pearson's correlation test. Data analysis was performed using the IBM SPSS Statistics 26 software package.

ELIGIBILITY:
Inclusion Criteria:

-Individuals aged 19-64 years

Exclusion Criteria:

* Individuals with physician-diagnosed psychological disorders.
* Individuals who regularly used medication or vitamin supplements.
* Individuals with alcohol or substance addiction.
* Pregnant or nursing women.

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample in Türkiye
Sampling Method: Non-Probability Sample
Enrollment: 498 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
My Nutrition Index | Baseline
  The My Nutrition Index (MNI), developed by Busgang et al. (2022), evaluates 34 dietary components, including fats, proteins, carbohydrates, vitamins, minerals, and electrolytes. The index is calculated based on 3-day food consumption records, considering factors like height, weight, gender, age, activity level, and lifestyle factors such as alcohol, smoking, and caffeine intake. MNI consists of four sub-dimensions: Macronutrient, Electrolyte, Vitamin, and Mineral Index, with scores ranging from 0 to 100, reflecting diet quality. The validity of the index was compared to the Healthy Eating Index-2015 (HEI-2015).
Healthy Eating Index-2015 | Baseline
  The Healthy Eating Index (HEI) was updated in 2015 and consists of 9 adequacy components: Whole Fruits, Total Fruits, Greens and Beans, Total Vegetables, Dairy, Whole Grains, Fatty Acids, Total Protein Foods, and Seafood and Plant Proteins, as well as 4 moderation components: Sodium, Refined Grains, Added Sugars, and Saturated Fats, resulting in a total of 13 components. HEI-2015 was calculated using the data obtained from the 3-day food consumption records of individuals. The index yields a minimum score of 0 and a maximum score of 100, with higher scores indicating better diet quality. Diet quality is categorized as follows: >80 represents good diet quality, 51-80 represents a diet quality that needs improvement, and ≤50 represents poor diet quality.

SECONDARY OUTCOMES:
International Physical Activity Questionnaire | Baseline
  In this study, the International Physical Activity Questionnaire Short Form (IPAQ) was utilized to determine the physical activity levels of the participants. The form, consisting of seven questions, provides information on sitting time, walking, moderately vigorous activities, and time spent in vigorous activities. The values obtained were evaluated according to the 'International Physical Activity Questionnaire Assessment Guide.' Based on this guideline, participants were classified into three categories: sedentary or less active, moderately active, and very active
Sociodemographic characteristics | Baseline
  Sociodemographic characteristics will be assessed using a structured questionnaire developed by the researchers. The questionnaire will include items measuring age, gender, education level, and income status. The results will be presented as numbers and percentages for each characteristic.
Body Mass Index (BMI) | Baseline
  Kilograms per square meter (kg/m2)
Body weight | Baseline
  Body weight in kg
Height | Baseline
  Height in cm

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No